CLINICAL TRIAL: NCT02710110
Title: The Impact of Respiratory Strength Training in Individuals With Amyotrophic Lateral Sclerosis (ALS)
Brief Title: Respiratory Strength Training in Persons With Amyotrophic Lateral Sclerosis (ALS)
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: ALS Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB201501172
Record Dates: First submitted 2016-02-26; First posted 2016-03-16 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Respiratory Physiological Phenomena; Capsaicin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active Respiratory Trainer (Experimental): Participants enrolled in this arm will be given the PowerLung trainer. The adjustable spring allows for discrete and calibrated changes to the valve, which in turn blocks air until sufficient inspiratory or expiratory pressure is applied by an individual. In addition, the Micro Mouth Pressure Meter, Pulmonary Function testing, videofluoroscopic swallowing study (VFSS), Swallowing Quality of Life Questionnaire (SWAL-QOL), Iowa Oral Pressure Instrument (IOPI), and capsaicin for use in the reflexive cough test.
  Interventions: Device: PowerLung trainer; Device: Micro Mouth Pressure Meter; Procedure: Pulmonary Function Testing; Procedure: Videofluoroscopic swallowing study; Other: Swallowing Quality of Life Questionnaire; Device: Iowa Oral Pressure Instrument; Drug: Capsaicin
- Sham Trainer (Sham Comparator): Participants enrolled in this arm will be given the PowerLung trainer; however, the adjustable spring allows for discrete and calibrated changes to the valve and these will not have any resistance. In addition, the Micro Mouth Pressure Meter, Pulmonary Function testing, videofluoroscopic swallowing study (VFSS), Swallowing Quality of Life Questionnaire (SWAL-QOL), Iowa Oral Pressure Instrument (IOPI), and capsaicin for use in the reflexive cough test.
  Interventions: Device: PowerLung trainer; Device: Micro Mouth Pressure Meter; Procedure: Pulmonary Function Testing; Procedure: Videofluoroscopic swallowing study; Other: Swallowing Quality of Life Questionnaire; Device: Iowa Oral Pressure Instrument; Drug: Capsaicin

INTERVENTIONS:
Device: PowerLung trainer — PowerLung trainer will be utilized which has both an inspiratory and expiratory loading capacity for training. A single daily training session will consist of three sets of 10 repetitions for a total of 30 inspiratory repetitions and 30 expiratory repetitions (i.e. 60 repetitions) for 5 days a week, for 3 months.
Device: Micro Mouth Pressure Meter — The participant will be seated with the nose occluded using a nose clip. After inhaling to total lung capacity, the participant will place his or her lips around the mouthpiece and blow out as forcefully as possible. A flange rubber mouthpiece will be used to overcome the inability of some individuals to create tight lip seal due to facial muscle weakness. Three trials will be performed and the patients highest Maximum Inspiratory Pressures (MIP) and Maximal Expiratory Pressure (MEP) used.
  Other Names: digital manometer; Micro Medical device
Procedure: Pulmonary Function Testing — Pulmonary Function testing will be performed using conventional methods and will include the following outcomes: forced vital capacity (FVC), sniff nasal inspiratory pressure (SNIP), peak expiratory flow (PEF), forced expiratory volume (FEV1) expressed as a percentage of predicted values.
Procedure: Videofluoroscopic swallowing study — Videofluoroscopic swallowing study will be performed to measure the oropharyngeal swallowing.
  Other Names: VFSS; X-ray of swallowing
Other: Swallowing Quality of Life Questionnaire — Swallowing Quality of Life Questionnaire (SWAL-QOL) will be used for participant reporting of swallow-related quality of life.
  Other Names: SWAL-QOL
Device: Iowa Oral Pressure Instrument — The IOPI is a device that measures the peak pressure performance of lingual strength and endurance via the action of a bulb placed on the hard palate.
  Other Names: IOPI
Drug: Capsaicin — A capsaicin challenge with three randomized blocks of 0, 50, 100, 200, and 500 μM capsaicin. The capsaicin will be dissolved in a vehicle solution consisting of 80% physiological saline, and 20% ethanol. Participants will be given the instruction "cough if you need to" prior to capsaicin delivery.The solution will be administered automatically upon detection of an inspired breath and there will be a minimum of one minute between each trial. This is to test the reflexive cough testing for upper airway sensitivity and motor thresholds.
  Other Names: Hot pepper

SUMMARY:
Dysphagia (swallow impairment), dystussia (cough impairment) and respiratory impairment are hallmark features of amyotrophic lateral sclerosis (ALS). These symptoms are the cause of fatal aspiration, malnutrition and respiratory insufficiency that together account for 91.4% of ALS mortality. Unfortunately, treatments to prolong and maintain these vital functions are currently lacking. Although the use of exercise in ALS is controversial, recent evidence suggests that mild to moderate intensity exercise applied early in the disease slows disease progression, improves motor function, preserves motor neuron number, reduces muscle hypoplasia, atrophy astrogliosis, and prolongs survival in animal models of ALS and human clinical trials.

This research study is designed to determine the impact of respiratory strength training on breathing, airway protection and swallowing in persons with Amyotrophic Lateral Sclerosis (ALS).

DETAILED DESCRIPTION:
This research study will measure the maximum inspiratory and expiratory pressure with secondary measures of respiration, swallow, cough, quality of life and global disease progression following twelve-weeks of treatment compared to the sham group.

As a participant two evaluations at the University of Florida Swallowing Systems Core laboratory located at Shands Hospital, Gainesville will take place. Each will take approximately two-hours and these will be spaced exactly three-months apart. During each evaluation tests will be performed to look at breathing, swallowing, and ability to cough doing standard clinical exams. In addition, some surveys about eating, speaking and quality of life will be taken.

Breathing Exercises: a home research therapist will train the participants how to use the hand-held respiratory trainer. Training for both treatment groups will be very similar, except the PowerLung trainer device will have an additional spring load valve inside it that will place a force on the respiratory muscles during training. The other breathing trainer will not have this spring so that no resistance will be placed on the respiratory muscles during training and this will represent an aerobic respiratory treatment. The breathing exercises will be completed five days a week for a total of three months (a total of 60 therapy sessions). During each session, a total of three sets of ten repetitions of breathing exercises will be performed. Once a week the home research therapist will visit and guide participants through the breathing exercise.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of probable or definite Amyotrophic Lateral Sclerosis (ALS),
* Amyotrophic Lateral Sclerosis Rating Scale Revised score greater than 34,
* forced vital capacity greater than 70%,
* cognition within normal limits as determined by Montreal assessment of cognition score >25

Exclusion Criteria:

* allergies to barium,
* tracheotomy or mechanical ventilation,
* diaphragmatic pacer,
* concurrent respiratory disease (e.g. COPD),
* pregnant at the time of the study due to radiation exposure

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2019-02-07 (Actual)

PRIMARY OUTCOMES:
Maximum Expiratory Pressure will be measured between the groups for a change from baseline to month 3 | Changes from baseline to month 3
  Maximum expiratory pressure is a measure of force generating capabilities as assessed by having subjects quickly inhale then rapidly blow out air into a handheld manometer (Micro Mouth Pressure Meter). Three trails will be performed and the highest will be used.
Maximum Inspiratory Pressure will be measured between the groups for a change from baseline to month 3 | Changes from baseline to month 3
  Maximum inspiratory pressure is a measure of force generating capabilities as assessed by having subjects quickly inhale then rapidly blow out air into a handheld manometer (Micro Mouth Pressure Meter). Three trails will be performed and the highest will be used.
Pulmonary function to measure the forced vital capacity (FVC) between the groups for a change from baseline to month 3 | Changes from baseline to month 3
  Pulmonary Function testing will be performed using a micro pressure meter. The participant will perform a maximum inhalation and then slowly blow out air into the mouthpiece of the meter. The following measurement will be displayed on the meter after the exhalation is complete forced vital capacity (FVC) expressed as a percentage of predicted values.
Sniff Nasal Inspiratory Pressure will be measured between the groups for a change from baseline to month 3 | Changes from baseline to month 3
Pulmonary function to measure the peak expiratory flow (PEF) will be measured between the groups for a change from baseline to month 3 | Changes from baseline to month 3
  Pulmonary Function testing will be performed using a micro pressure meter. The participant will perform a maximum inhalation and then slowly blow out air into the mouthpiece of the meter. The following measurement will be displayed on the meter after the exhalation is complete peak expiratory flow (PEF) expressed as a percentage of predicted values.
Pulmonary function to measure the forced expiratory volume (FEV1) will be measured between the groups for a change from baseline to month 3 | Changes from baseline to month 3
  Pulmonary Function testing will be performed using a micro pressure meter. The participant will perform a maximum inhalation and then slowly blow out air into the mouthpiece of the meter. The following measurement will be displayed on the meter after the exhalation is complete forced expiratory volume (FEV1) expressed as a percentage of predicted values.

SECONDARY OUTCOMES:
The Penetration-aspiration scale will be used to measure swallowing function | Changes from baseline to month 3
  Videofluoroscopic swallowing study will be performed to measure the oropharyngeal swallowing.
Lingual strength will be measured between the groups for a change from baseline to month 3 | Changes from baseline to month 3
  The Iowa Oral Pressure Instrument device will measure the peak performance of lingual strength a via the action of a bulb placed on the hard palate. To assess maximum anterior isometric pressure, the bulb will be placed on the roof of the mouth and the participant will raise his or her tongue to apply pressure to this bulb and then quickly release the tongue back into a neutral position. This repetitive tongue movement will be performed three times and values will be recorded.
Lingual endurance will be measured between the groups for a change from baseline to month 3 | Changes from baseline to month 3
  The Iowa Oral Pressure Instrument device will measure the peak performance of maximum lingual endurance time by instructing the participant to place the bulb on the roof of the mouth and then apply and sustain pressure to the bulb for as long as he/she can at a threshold of 20% of the maximum anterior isometric pressure. The maximum lingual endurance time will also be recorded.
Voluntary cough function will be measured between the groups for a change from baseline to month 3 | Changes from baseline to month 3
  Voluntary cough function will be assessed using an oral pneumotachograph, connected to a spirometer filter during voluntary cough production. The participant will be seated with a respiratory face-mask held in place by the examiner and instructed to complete three tidal breaths into the face-mask, airflow signal will be measured
Reflexive cough will be measured between the groups for a change from baseline to month 3 | Changes from baseline to month 3
  Reflexive cough will be assessed using an oral pneumotachograph, differential pressure transducer, and have a side port with a one-way inspiratory valve for nebulizer connection. The nebulizer will deliver three randomized blocks of 0, 50, 100, 200, and 500 μM capsaicin.

CONTACTS AND LOCATIONS:
Overall Officials: Emily K Plowman, Ph.D., Principal Investigator — University of Florida
Locations (1):
- UF Health Shands, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No